CLINICAL TRIAL: NCT05452681
Title: Piloting Y-AMBIENT: A Quality of Life Intervention for Young African American Breast Cancer Survivors
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Timiya Nolan, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: IRB-300012133
Record Dates: First submitted 2022-07-06; First posted 2022-07-11 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer; Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Y-AMBIENT (Experimental): Y-AMBIENT is a four-month, telephone-based intervention that includes three themed education sessions with three follow-up sessions, written materials, and videos. All themed education and follow-up sessions are conducted according to the respective Y-AMBIENT session outlines and audio-recorded. Session 1, titled "My Self, My Soul," covers topics related to spiritual growth and finding meaning in illness. Session 2, titled "My Body," covers topics related to breast changes, aches/pains, fatigue, and weight changes. Session 3, titled "My Mind and My Relationships," covers topics related to anxiety, fear, and relationships with others. The sessions will take approximately one hour, with follow-ups lasting about 20 minutes. Participants will receive both printed and electronic PDF versions of written materials, in addition to video links, to reinforce content delivered during Sessions.
  Interventions: Other: Educational Intervention; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Attention Control (Active Comparator): The control condition will consist of receiving a culturally-targeted cookbook applied by an adapted "Food for Thought" cookbook, a guide to grocery shopping smart, and telephone socialization calls. We opted to use the cookbook and guide as conversation pieces given cultural practices associated with food and avert financial constraints with shopping tips. During three, one-hour socialization calls, we will use scripted questions to encourage discussion about the participant, cookbook and guide, and obtain information about survivorship concerns without providing coaching. The follow-up calls will last about 20 minutes.
  Interventions: Other: Quality-of-Life Assessment; Other: Questionnaire Administration; Other: Control Intervention

INTERVENTIONS:
Other: Educational Intervention — Receive Y-AMBIENT
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Y-AMBIENT
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies
Other: Control Intervention — Receive cookbook and socialization calls
  Other Names: Attention control intervention; Control Intervention, Attention
  Arms: Attention Control

SUMMARY:
The purpose of this two-arm pilot RCT is to evaluate processes and preliminary outcomes of a targeted QOL intervention vs. an attention control among young AA survivors post-treatment for early (I-II) & late (III) stage breast cancer.

DETAILED DESCRIPTION:
Primary Objectives

I. Evaluate feasibility and acceptability of Y-AMBIENT and an attention control among young African American breast cancer survivors.

II. Explore the degree to which the Y-AMBIENT vs. attention control affects preliminary health-related outcomes among young African American (AA) survivors.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I (Y-AMBIENT): Patients receive three themed education sessions over 1 hour each, written materials, and videos at month 1. Patients also participate in 3, 20 minutes telephone reinforcement calls to discuss how they are doing and discuss any concerns that they are still managing at months 2, 3, and 4.

ARM II (ATTENTION CONTROL): Patients receive three themed education sessions over 1 hour each, written materials, and videos at month 1. Patients also participate in 3, 20 minutes telephone reinforcement calls to discuss how they are doing and discuss any concerns that they are still managing at months 2, 3, and 4.

After completion of study, patients are followed up at 1 month.

ELIGIBILITY:
Inclusion Criteria:

* Biologically born women
* Self-identify as AA
* Are aged 18 to 44 years on study entry
* Are diagnosed with breast cancer stage I-III
* Have completed treatment with chemotherapy and/or radiation for stage I-III breast cancer prior to study entry
* Are English- speaking
* Have telephone and internet access

Exclusion Criteria:

* Participation in formal survivorship navigation programs because they are associated with improved health- related outcomes, which could be a confounder

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of screen-eligible patients enrolled by consent | Up to 2 years
  Descriptive statistics will be used to compute the proportion of screen-eligible patients enrolled by consent. Proportions will be computed, along with 95% confidence intervals, to indicate the precision of the point estimate.
Proportion of patients that complete all (five) study contacts of intervention | Up to 2 years
  Descriptive statistics will be used to compute proportion of patients that complete all (five) study contacts of the intervention. Proportions will be computed, along with 95% confidence intervals, to indicate the precision of the point estimate.
Acceptability/Relevance of Intervention Sessions | Up to 2 years
  Will use qualitative interview to assess participants' perceptions of its acceptability/relevance of each of the six study contacts, using a Likert scale 0 to 10 with 0 being not at all satisfied/useful and 10 being completely satisfied/useful and an open ended question to understand why each score was provided. A composite score will be determined, where higher scores equate to higher acceptability/relevance. Descriptive statistics will be computed, along with 95% confidence intervals, to indicate the precision of the point estimate. Qualitative responses will be analyzed for content.
Participation in aspects of protocol | Up to 2 years
  Will use qualitative interview to assess participants' engagement by review of task completion to participate in aspects of the protocol (as an indicator of participant burden). There are a total of six sessions to complete and seven videos to review. Descriptive statistics will be used to compute the proportion of participant self-reported effectiveness of each intervention via the logs. Completion of tasks indicates greater willingness to participate.
Use of proposed self-management strategies and perceived effectiveness | Up to 2 years
  Will use qualitative interview to assess participants' engagement by review of use of proposed self-management strategies and their perceived effect on quality of life concerns using a Likert scale 0 to 10 with 0 being not at all effective and 10 being most effective. Descriptive statistics will be used to compute the proportion of participant self-reported effectiveness of each intervention via the logs. Qualitative responses will be analyzed for content.
Medical Outcomes Survey Short-Form (SF-36) | Baseline up to 1 month post-intervention
  The SF-36 is a well-established measure of health status in cancer survivors. SF-36 includes one multi-item scale assessing eight health concepts: limitations in physical activity, social activity, role activity, bodily pain, psychological distress, limitations in social activity due to emotional distress, vitality, and general health perceptions. The scale ranges from 0-100. Higher scores indicate better functioning.
  Will use mixed-effects linear modeling for repeated measures to (a) test the fixed effect of time, intervention group, and their interaction; (b) derive within-group and between-group contrast estimates on the change from baseline at each follow-up.
PROMIS Global Health10 | Baseline up to 1 month post-intervention
  The PROMIS Global Health 10 is a well-established measure of health status in cancer survivors. It assesses health and functioning including overall physical health, mental health, social health, pain, fatigue, and overall perceived quality of life. Higher scores indicate better functioning.
  Will use mixed-effects linear modeling for repeated measures to (a) test the fixed effect of time, intervention group, and their interaction; (b) derive within-group and between-group contrast estimates on the change from baseline at each follow-up.
(Functional Assessment of Chronic Illness Therapy Spiritual Well-Being (FACT-Sp 12) | Baseline up to 1 month post-intervention
  The FACIT-SP-12 is the most widely used measure of spiritual well-being among those with cancer. Its subscales measure faith, meaning, and peace. Higher scores reflect higher well-being.
  Will use mixed-effects linear modeling for repeated measures to (a) test the fixed effect of time, intervention group, and their interaction; (b) derive within-group and between-group contrast estimates on the change from baseline at each follow-up.
MOS Modified Social Support Survey | Baseline up to 1 month post-intervention
  MOS assesses dimensions of social support with four functional support scales: emotional/informational, tangible, affectionate, and positive social interaction. The scale ranges from 0-100. Higher scores indicate greater social support.
  Will use mixed-effects linear modeling for repeated measures to (a) test the fixed effect of time, intervention group, and their interaction; (b) derive within-group and between-group contrast estimates on the change from baseline at each follow-up.
PROMIS Applied Cognition - General Concerns short form (8- item) | Baseline up to 1 month post-intervention
  This instrument measures working memory, speed of processing, and executive control of cognitive functioning. Higher scores reflect higher perceived cognitive functionality.
  Will use mixed-effects linear modeling for repeated measures to (a) test the fixed effect of time, intervention group, and their interaction; (b) derive within-group and between-group contrast estimates on the change from baseline at each follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Timiya Nolan, PhD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No